CLINICAL TRIAL: NCT07268482
Title: Randomised Control Study of Using a Pressure Monitoring Technology for Improving the Targeted Application, Monitoring, and Maintenance of Compression Therapy in Patients With Venous Leg Ulcers
Brief Title: Assessing Sensor-Guided Compression Therapy for Venous Leg Ulcers Healing Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Feeltect Limited (Industry)
Collaborators: University of Galway (Other); CORRIB-CURAM Vascular Group, University of Galway, Galway, Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MERLIN251112WoundCompress
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Venous Leg Ulcer (VLU)
Keywords: Venous Leg Ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive standard care and use the pressure-sensing device with a blinded application (no feedback provided), with data transmitted for monitoring.
- Treatment (Experimental): The treatment group will also receive the same standard care, with the same type of compression bandages, but use the device with real-time feedback, enabling nurses to apply the targeted pressure reliably, and patients and carers to monitor pressure trends and apply additional compression as needed.
  Interventions: Device: A connected-health, pressure-sensing system for monitoring sub-bandage pressure during compression therapy

INTERVENTIONS:
Device: A connected-health, pressure-sensing system for monitoring sub-bandage pressure during compression therapy — The study will be conducted at merlin Park University Hospital Galway and will include two cohorts: a control group receiving standard unguided compression therapy with blinded device use (i.e. compression pressures will be blinded at the point of care but monitored remotely), and an intervention group using Tight Alright technology to guide compression application and reapplication. Outcomes will include wound healing rates, time to healing, pressure maintenance, patient adherence, and usability. The study aims to determine whether integrating connected-health pressure monitoring can improve consistency of compression therapy, accelerate healing, and enhance patient engagement in the treatment of venous leg ulcers
  Arms: Treatment

SUMMARY:
The investigators are conducting a study to find out if a new system can help improve the care of people with venous leg ulcers (VLU). Venous leg ulcers are wounds on the lower leg that need compression bandages to help them heal.

In this study, patients will be randomly placed into one of two groups:

* Group 1: Will receive the usual care for VLUs.
* Group 2: Will use a new connected health system, called Tight Alright, along with their usual care.

The Tight Alright system includes a small, wearable device that sits under a patient's bandage. This device measures the pressure at three points on the patient's lower leg and sends the information wirelessly to a mobile app. The app shows real-time pressure readings and also sends the data to a secure cloud database. This allows the patient's healthcare team to monitor their bandage pressure remotely and make sure it is just right.

The aim is to help nurses and doctors apply the correct pressure every time, which is important for healing. The system can also alert the patient's healthcare team if the pressure drops, so they can decide if a patient's bandage needs adjusting, even when the patient is at home.

The investigators will follow all participants for 90 days and then compare how well the ulcers have healed in both groups. This will help us find out if the new system can improve healing and make treatment safer and more effective.

DETAILED DESCRIPTION:
This proposed study is a prospective, randomized, controlled trial designed to evaluate the effectiveness of a pressure-sensing compression therapy device for VLUs. Eligible patients will be identified through a combination of ankle brachial index measurements, venous duplex ultrasound, comprehensive wound assessment, and a review of their care plans. Informal carers, such as family members or friends, may participate to assist with device use and data transmission. All participants will receive detailed study information and provide written informed consent prior to enrolment.

After enrolment, each patient will enter a two-week run-in period during which they will receive standard care. During this time, their wound will be photographed and measured using eKare wound monitoring technology. Patients whose wounds decrease in size by more than 40% during this period will be excluded to maintain a homogeneous study population. All participants will receive thorough training on device usage and data transmission, with their proficiency evaluated prior to the start of the study. Those who meet the inclusion criteria will then be randomly assigned to either the control or treatment group according to a computer-generated allocation schedule.

The control group will receive standard care and use the pressure-sensing device with a blinded application (no feedback provided), with data transmitted for monitoring.

The treatment group will also receive the same standard care, with the same type of compression bandages, when possible, but use the device with real-time feedback, enabling nurses to apply the targeted pressure reliably, and patients and carers to monitor pressure trends and apply additional compression as needed.

Throughout 90 days all patients will continue with scheduled wound care, and at each visit, compression pressures and wound area will be assessed. Patients will take the device home, transmit daily pressure readings, and be instructed to apply additional compression if pressures fall below target thresholds. Study nurses will monitor data remotely and provide follow-up as needed. A quality-of-life questionnaire will also be given to the patients to fill in every two weeks.

Patients will exit the study after 90 days, upon wound healing, or if complications arise. A final clinic evaluation and discharge questionnaire will be completed to assess patient experience and technology usability.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic venous leg ulcers (≥6-week and ≤5-year durations) currently in compression therapy treatment.
* Between 5 and 100 cm2 wound area at randomization.
* Ankle brachial pressure index (ABPI) of >0,8
* Capable of using use a smart device.

Exclusion Criteria:

* Uncontrolled diabetes [haemoglobin A1c (HbA1c) ≥12% in the last 3 months]
* Index ulcer has active infection on day of inclusion requiring systemic antibiotic therapy
* Renal failure
* Exposed tendon, ligament, muscle or bone in the index ulcer
* Osteomyelitis, cellulitis or gangrene in study limb
* Subjects with an amputation above transmetatarsal in study limb
* Active malignancy affecting study limb
* Index ulcer is of arterial aetiology (ABPI <0.8)
* Pregnant or breast-feeding women or women of childbearing potential not willing to use a method of highly effective contraception for the duration of the study
* Planned vascular surgery, angioplasty or thrombolysis procedures during study period. Or patients who are within six weeks of having had such a procedure
* Planned surgical procedure during study period for the index wound
* Prior skin replacement, negative-pressure therapy and ultrasound therapy to the study wound in the two weeks before screening
* Currently receiving or has received radio or chemotherapy within three months of randomisation
* Index wound would require ultrasound near an electronic implant or prosthesis
* Not capable of providing informed consent
* Currently enrolled in or has been enrolled in another investigation device or drug trial in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Percentage area reduction per day | From enrollment to the end of treatment 9 months
  The weekly rate of wound area reduction (cm2) represented as a percentage, calculated by comparing the wound size at the end of the treatment (Aend) with the wound size at the start of treatment (Astart) and normalising for the length of time for treatment (T). (Aend - Astart)/Astart*100/T

SECONDARY OUTCOMES:
Average pressure applied to each patient | From enrolment to the end of treatment 9 months
  Tight Alright enables accurate real-time measurement of sub-bandage compression pressure (in mmHg). This outcome will measure the average pressure applied over the duration of treatment
Percentage of patients healed | From enrolment to the end of treatment 9 months
  The percentage of patients healed completely within the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Merlin Park University Hospital, Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No